



## STATISTICAL ANALYSIS PLAN

Project Number: GLPG0634

Study Number: GS-US-419-3896 (GLPG0634-CL-310)

Study Title: A Long-Term Extension Study to Evaluate the Safety of Filgotinib in

Subjects with Crohn's Disease

Development Phase: 3

Status: Final

Version: 2.0 Date: 1-Aug-2023

EudraCT: 2016-002763-34 IND: 129646

Sponsor: Galapagos NV, Generaal De

Wittelaan L11 A3, 2800 Mechelen, Belgium

Biostatistician:

Medical Leader:

#### **Confidentiality Statement**

The information contained in this document is privileged and confidential. It is the property of Galapagos NV and may not be used, disclosed, reproduced or otherwise disseminated within your organization or communicated to any third parties without the express written authorization of Galapagos NV.

## TABLE OF CONTENTS

| TA | BLE OF | CONTENTS | 2 |
|---|---|---|---|
| LIS | T OF A | BBREVIATIONS | 5 |
| 1. | INTR | ODUCTION | 7 |
| | 1.1. | Study Objectives | |
| | 1.2. | Study Design | |
| | 1.3. | Sample Size and Power | |
| 2. | TYPE | OF PLANNED ANALYSIS | 9 |
| | 2.1. | Interim Analyses | 0 |
| | 2.2. | Final Analysis | |
| 3. | GENERAL CONSIDERATIONS FOR DATA ANALYSES | | |
| | 3.1. | 3.1. Analysis Sets | |
| | | 3.1.1. All Enrolled Analysis Set | |
| | | 3.1.2. Safety Analysis Set | 10 |
| | 2.2 | | |
| | 3.2. | Subject Grouping | |
| | 3.3.<br>3.4. | Strata and Covariates | |
| | 3.5. | Multiple Comparisons | |
| | 3.6. | Missing Data and Outliers | |
| | | 3.6.1. Missing Data | |
| | | 3.6.2. Outliers | |
| | 3.7. | Data Handling Conventions and Transformations | |
| | 3.8. | Analysis Visit Windows | |
| | | 3.8.1. Definition of Study Day | |
| | | 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Visit | 13 |
| | | Window | 16 |
| | | 3.8.4. Definition of Baseline | 16 |
| 4. | SUBJ | ECT DISPOSITION | 17 |
| | 4.1. | Subject Enrollment and Disposition | 17 |
| | 4.2. | Extent of Study Drug Exposure and Adherence | |
| | | 4.2.1. Duration of Exposure to Study Drug | |
| | | 4.2.2. Adherence to Study Drug | |
| | | 4.2.2.1. On-Treatment Adherence | |
| | 4.3. | Protocol Deviations | |
| | 4.4. | Assessment of COVID-19 (Coronavirus Disease 2019) and Ukrainian Conflict Impact | |
| | | 4.4.1. Study Drug or Study Discontinuation | |
| | | 4.4.2. Study Drug Interruption | |
| | | 4.4.4. Missed or Virtual Visits | |
| | | 4.4.5. Adverse Events. | |
| | | 4.4.6. Comments | |
| 5. | BASE | LINE CHARACTERISTICS | 22 |
| | 5.1. | Demographics and Baseline Characteristics | 22 |
| | 5.2. | Other Baseline Characteristics | |
| | 5.3. | Medical History | |
| 6. | FFFI | CACY ANALYSES | |
| υ. | U. EFFICACT ANALIBES | | |

| | 6.1. | | | | |
|---|---|---|---|---|---|
| | | 6.1.1. | | OAI and PRO2 Scores | |
| | 6.2. | | | DCC D 1 '4 | |
| | | 6.2.1. | | Efficacy Endpoints | |
| | 6.2 | 6.2.2. | | fficacy Endpoints | |
| | 6.3. | Subgrou | Analyses | | 23 |
| | 6.5. | | _ | fied Efficacy Analyses | |
| 7. | SAFE | TY ANAI | YSES | | 29 |
| | 7.1. | Adverse | | | |
| | | 7.1.1. | | ctionary | |
| | | 7.1.2. | | verity | |
| | | 7.1.3. | | dverse Events to Study Drug | |
| | | 7.1.4. | | th Study Drug | |
| | | 7.1.5. | Serious Adverse I | Events | 29 |
| | | 7.1.6. | | ent Adverse Events | |
| | | | 7.1.6.1. Defi | nition of Treatment-Emergent Adverse Events | 30 |
| | | | 7.1.6.2. Inco | mplete Dates | 30 |
| | | 7.1.7. | | verse Events and Deaths | 30 |
| | | | | maries of AE incidence in Combined Severity Grade<br>sets | 30 |
| | | 7.1.8. | Adverse Events o | f Interest | 32 |
| | | | | diovascular Safety Endpoint Adjudication Committee | |
| | 7.2. | Laborate | | | |
| | | 7.2.1. | | meric Laboratory Results | |
| | | 7.2.2. | Graded Laborator | y Values | 35 |
| | | | | atment-Emergent Laboratory Abnormalities | |
| | | | | ntment-Emergent Marked Laboratory Abnormalities | |
| | | | 7.2.2.3. Sum | maries of Laboratory Abnormalities | 35 |
| | | 7.2.3. | | poratory Evaluations | |
| | 7.3. | Body W | | 3 | |
| | 7.4. | Concom | tant Medications | | 37 |
| | 7.5. | Electroc | ardiogram Results | | 38 |
| | 7.6. | Other Sa | fety Measures | | 38 |
| 9. | SOFT | WARE | | | 40 |
| 10. | SAP I | REVISION | | | 41 |
| 11. | APPE | NDICES . | | | 43 |

## LIST OF IN-TEXT TABLES

| Table 3-1. | Analysis Visit Windows for CDAI, PRO2, Vital Signs, Weight, Hematology and Chemistry | 13 |
|---|---|---|
| Table 3-2. | Analysis Visit Windows for Lipid Profile, Serum Immunoglobulin | |
| | | 15 |
| Table 11-1. | Calculation of Total CDAI Score | 47 |
| Table 11-2. | Calculation of PRO2 Components | |
| Table 11-3. | Calculation of CDAI Patient-Reported Outcome Components and PRO2 Scores for | |
| | Baseline and Post-baseline Visits | 49 |
| Table 11-4. | Sources of Information for Calculating CDAI and PRO2 Scores | 50 |
| Table 11-5. | Example Search Terms for "COVID-19" and "Virtual" Used to Identify | |
| | Missed/Virtual Visits | 51 |
| | LIST OF IN-TEXT FIGURES | |
| Figure 1 | Selection of Diary Data for the Calculation for Baseline and Postbaseline Visits | 49 |

#### LIST OF ABBREVIATIONS

AE adverse event

AEI adverse events of interest
ALT alanine aminotransferase
AST aspartate aminotransferase

ASTE arterial systemic thromboembolism

BMI body mass index CD Crohn's disease

CDAI Crohn's Disease Activity Index

CI confidence interval

COVID-19 coronavirus disease 2019

CRF case report form
CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

CV cardiovascular

CVEAC cardiovascular safety endpoint adjudication committee

DMC data monitoring committee

ECG electrocardiogram

eCRF electronic case report form

ET early termination
Hb hemoglobin

HDL high-density lipoprotein
HLGT high-level group term
HLT high-level term

ID identification

Ig immunoglobulin

LDL low-density lipoprotein
LOQ limit of quantitation
LTE long term extension
LTT lower-level term

MACE major adverse cardiovascular events

MedDRA Medical Dictionary for Regulatory Activities

MI myocardial infarction

MST MedDRA search term

NLP Natural Language Processing

GS-US-419-3896 (GLPG0634-CL-310)

| PRO2 | natient renor | ted outcome c | onsisting o | f 2 items: | abdominal | pain severity | v and liquid stool |
|---|---|---|---|---|---|---|---|
| 1102 | patient repor | ica cateonie c | onoibung o | 1 2 Itellio. | acaciiiiiai | pulli be verit | y und niquid bloom |

frequency

PT preferred term
PTx post-treatment
Q1 first quartile
Q3 third quartile

SAE serious adverse event
SAP statistical analysis plan
SD standard deviation
SE standard error

SMQ Standardized MedDRA Query

SOC system organ class
TE treatment-emergent

TEAE treatment-emergent adverse event

TFLs tables, figures, and listings ULN upper limit of normal

V-Day visit day

VAS Visual Analogue Scale
VTE venous thromboembolism
WHO World Health Organization

#### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis methods and data presentations to be used in tables, figures, and listings (TFLs) in the interim analyses and clinical study report (CSR) for Study GS-US-419-3896 (GLPG0634-CL-310). This SAP is based on the study protocol Amendment 8 dated 2 December 2021 and the electronic case report form (eCRF). The SAP will be finalized before unblinding of Study GS-US-419-3895 (GLPG0634-CL-309), at which time this study will be unblinded. Any changes made after the finalization of the SAP will be documented in the CSR.

#### 1.1. Study Objectives

The primary objective of this study is:

 To observe the long-term safety of filgotinib in subjects who have completed or met protocol specified efficacy discontinuation criteria in a prior filgotinib treatment study for Crohn's disease (CD)

The secondary objective of this study is:

 To evaluate the effect of filgotinib on Patient Reported Outcomes (PRO2) and Crohn's Disease Activity Index (CDAI) scores

#### 1.2. Study Design

This is a long-term extension (LTE) study to evaluate the safety of filgotinib administered to subjects with CD. Some subjects will receive open-label drug and some will continue to receive the blinded study drug assigned in the parent study until subject's treatment in the corresponding parent study (GS-US-419-4015, GS-US-419-4016, or GS-US-419-3895) is unblinded. The duration of treatment is up to 432 weeks.

In general, subjects who fully complete a parent study blinded will continue blinded treatment at the same regimen in the present study on 200 mg filgotinib, 100 mg filgotinib, or placebo. Subjects who enroll from a parent study and receive blinded treatment in the GS-US-419-3896 study will have their GS-US-419-3896 treatment assignment unblinded when the parent study is unblinded. After the study unblinding, subjects will continue on the same dose of open-label filgotinib as they had been receiving in blinded treatment; whereas subjects on placebo treatment

will discontinue study drug and study participation. Subjects who exit a parent study due to disease worsening or failure to meet response or remission criteria will receive open-label 200 mg filgotinib, with the exception of US and Korea males in this category who were not considered biologic refractory who will receive open-label 100 mg filgotinib.

This study includes:

- Day 1
- Treatment Visits: Week 2, Week 4, Week 12, and then every 12 weeks thereafter
- Post-Treatment (PTx) safety assessments (30 days after the last dose of study drug) for subjects who complete all study treatment visits or discontinue early

For additional details, please see the Schedule of Assessments in Appendix 1.

### 1.3. Sample Size and Power

No formal hypothesis testing is planned for this study and sample size calculation is not conducted. All subjects who have completed or met protocol-specified efficacy discontinuation criteria in a parent study (GS-US-419-4015, GS-US-419-4016, or GS-US-419-3895) may enroll in this study. The projected number of subjects enrolled is approximately 1000.

## 2. TYPE OF PLANNED ANALYSIS

## 2.1. Interim Analyses

Prior to the final analysis, interim analyses may be performed for regulatory submission and/or for publication purposes. The first interim analysis is planned to align with the final analysis of Study GS-US-419-3895, at which time this study will be unblinded.

Interim analyses may present a subset of the analyses included in this analysis plan.

## 2.2. Final Analysis

The final analysis will be performed after all subjects have completed the study.

#### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

All analyses described in this SAP will include data from the LTE study (GS-US-419-3896) exclusively, not from the corresponding parent studies, except for subgroup analyses based on parent study completion status. Consequently, any reference to study drug (e.g., first dosing date) implies study drug administered in Study GS-US-419-3896, unless specifically stated otherwise.

Analysis results will be presented using descriptive statistics. For categorical variables, the number and percentage of subjects in each category will be presented; for continuous variables, the number of subjects (n), mean, standard deviation (SD) or standard error (SE), median, first quartile (Q1), third quartile (Q3), minimum, and maximum will be presented.

By-subject listings will be presented for all subjects in the All Enrolled Analysis Set and sorted by subject identification (ID) number, visit date, and time (if applicable). Data collected on log forms, such as adverse events (AEs), will be presented in chronological order within the subject. The treatment group to which subjects were assigned at enrollment will be used in the listings. Age (on the first dosing day in the LTE), sex at birth, race, and ethnicity will be included in the listings, as space permits.

#### 3.1. Analysis Sets

Analysis sets define the subjects to be included in an analysis. Analysis sets and their definitions are provided in this section. The analysis set will be identified and included as a subtitle of each table, figure, and listing.

For each analysis set, the number and percentage of subjects eligible for inclusion, as well as the number and percentage of subjects who were excluded and the reasons for their exclusion (if available), will be summarized by treatment group.

A listing of reasons for exclusion from analysis sets (if applicable) will be provided by subject.

#### 3.1.1. All Enrolled Analysis Set

All Enrolled Analysis Set includes all subjects who enrolled into this study as recorded in the Enrollment eCRF.

#### 3.1.2. Safety Analysis Set

The Safety Analysis Set includes all subjects who took at least 1 dose of study drug in Study GS-US-419-3896. This is the primary analysis set for safety and efficacy analyses.

#### 3.1.3.

#### 3.2. Subject Grouping

For analyses based on the Safety Analysis Set and grouped according to the actual treatment received. The actual treatment received will differ from the assigned treatment only when their actual treatment differs from assigned treatment for the entire treatment duration.

For analyses of baseline characteristics and efficacy endpoints in the subset of subjects who rolled over into the LTE due to failure to meet response/remission criteria at W10 (see Section 3.4 and Section 6.3), subjects will be grouped according to the actual treatment received in both the parent study and the LTE study.

#### 3.3. Strata and Covariates

This study does not use a stratified randomization schedule when enrolling subjects. No covariates will be included in safety and efficacy analyses.

#### 3.4. Subgroup Analyses

Subgroup analyses will be performed for the group of subjects who rolled over into the LTE due to failure to meet response/remission criteria at W10 (induction non-responders):

- Overall, and,
- O By number of prior exposures to biologic agent (0 vs  $\geq$ 1).

Subgroup analyses for efficacy endpoints are specified in Section 6.3.

#### 3.5. Multiple Comparisons

Adjustments for multiplicity will not be made, because no formal statistical testing will be performed in this study.

#### 3.6. Missing Data and Outliers

### 3.6.1. Missing Data

In general, missing data will not be imputed unless methods for handling missing data are specified. Exceptions are presented in this document.

For missing last dosing date of study drug, imputation rules are described in Section 4.2. Imputation and calculation rules for missing patient diary data are described in Section 6.1. The handling of missing or incomplete dates for AE onset is described in Section 7.1.6.2, and for concomitant medications in Section 7.4.

#### **3.6.2. Outliers**

Outliers will be identified during the data management and data analysis process, but no sensitivity analyses will be conducted. All data, including outliers, will be included in the data analysis, unless otherwise specified.

## 3.7. Data Handling Conventions and Transformations

In general, age (in years) on the date of the first dose of study drug will be used for analyses and presented in listings. If an enrolled subject was not dosed with any study drug, the enrollment date will be used instead of the first dosing date of study drug. If only the birth year is collected on the CRF, "01 July" will be used for the unknown birth day and month for the purpose of age calculation. If only birth year and month are collected, "15" will be used for the unknown birth day.

Non-pharmacokinetic data that are continuous in nature but are less than the lower limit of quantitation (LOQ) or above the upper LOQ will be imputed as follows:

- A value that is 1 unit less than the lower LOQ at the same precision level of the originally reported value will be used to calculate descriptive statistics if the datum is reported in the form of "< x" (where x is considered the lower LOQ). For example, if the values are reported as < 50 and < 5.0, values of 49 and 4.9, respectively, will be used to calculate summary statistics. An exception to this rule is any value reported as < 1 or < 0.1, etc. For values reported as < 1 or < 0.1, a value of 0.9 or 0.09, respectively, will be used to calculate summary statistics.
- A value that is 1 unit above the upper LOQ will be used to calculate descriptive statistics if the datum is reported in the form of "> x" (where x is considered the upper LOQ). Values with decimal points will follow the same logic as above.
- The lower or upper LOQ will be used to calculate descriptive statistics if the datum is reported in the form of " $\leq$  x" or " $\geq$  x" (where x is considered the lower or upper LOQ, respectively).

## 3.8. Analysis Visit Windows

#### 3.8.1. Definition of Study Day

The First Dosing Date is defined as the date when subjects take the first dose of study drug in this study, as recorded in the Study Drug Administration eCRF.

The Last Dosing Date is defined as the date when subjects take the last dose of study drug in this study, as recorded in the Study Drug Administration eCRF.

Study day will be calculated from the first dosing date of study drug and derived as follows:

- For days on or after the first dosing date: Assessment Date First Dosing Date + 1
- For days prior to the first dosing date: Assessment Date First Dosing Date

Therefore, Study Day 1 is the day of first dose of study drug administration.

Baseline is defined as the last available observation on or prior to the first dosing date, unless otherwise specified.

#### 3.8.2. Analysis Visit Windows

Subject visits might not occur on protocol-specified days. Therefore, for the purpose of analysis, observations will be assigned to analysis windows.

The analysis windows for CDAI, PRO2, vital signs, weight, hematology, and chemistry are provided in Table 3-1. The analysis windows for lipid profile, serum immunoglobulin, re provided in Table 3-2. The analysis windows for

Table 3-1. Analysis Visit Windows for CDAI, PRO2, Vital Signs, Weight, Hematology and Chemistry

| | | Visit Window Study Day | |
|---------------|-------------------|------------------------|-------------|
| Nominal Visit | Nominal Study Day | Lower Limit | Upper Limit |
| Baseline | 1 | (none) | 1 |
| Week 2 | 15 | 2 | 22 |
| Week 4 | 29 | 23 | 57 |
| Week 12 | 85 | 58 | 127 |
| Week 24 | 169 | 128 | 211 |
| Week 36 | 253 | 212 | 295 |
| Week 48 | 337 | 296 | 379 |
| Week 60 | 421 | 380 | 463 |
| Week 72 | 505 | 464 | 547 |
| Week 84 | 589 | 548 | 631 |
| Week 96 | 673 | 632 | 715 |
| Week 108 | 757 | 716 | 799 |
| Week 120 | 841 | 800 | 883 |

| | | Visit Window Study Day | |
|---------------|-------------------|------------------------|-------------|
| Nominal Visit | Nominal Study Day | Lower Limit | Upper Limit |
| Week 132 | 925 | 884 | 967 |
| Week 144 | 1009 | 968 | 1051 |
| Week 156 | 1093 | 1052 | 1135 |
| Week 168 | 1177 | 1136 | 1219 |
| Week 180 | 1261 | 1220 | 1303 |
| Week 192 | 1345 | 1304 | 1387 |
| Week 204 | 1429 | 1388 | 1471 |
| Week 216 | 1513 | 1472 | 1555 |
| Week 228 | 1597 | 1556 | 1639 |
| Week 240 | 1681 | 1640 | 1723 |
| Week 252 | 1765 | 1724 | 1807 |
| Week 264 | 1849 | 1808 | 1891 |
| Week 276 | 1933 | 1892 | 1975 |
| Week 288 | 2017 | 1976 | 2059 |
| Week 300 | 2101 | 2060 | 2143 |
| Week 312 | 2185 | 2144 | 2227 |
| Week 324 | 2269 | 2228 | 2311 |
| Week 336 | 2353 | 2312 | 2395 |
| Week 348 | 2437 | 2396 | 2479 |
| Week 360 | 2521 | 2480 | 2563 |
| Week 372 | 2605 | 2564 | 2647 |
| Week 384 | 2689 | 2648 | 2731 |
| Week 396 | 2773 | 2732 | 2815 |
| Week 408 | 2857 | 2816 | 2899 |
| Week 420 | 2941 | 2900 | 2983 |
| Week 432 | 3025 | 2984 | ≥ 3025 |

CDAI = Crohn's Disease Activity Index; PRO2 = patient reported outcome consisting of 2 items: abdominal pain severity and liquid stool frequency

Analysis Visit Windows for Lipid Profile, Serum Immunoglobulin, **Table 3-2.** 

| | | Visit Window Study Day | |
|---------------|-------------------|------------------------|-------------|
| Nominal Visit | Nominal Study Day | Lower Limit | Upper Limit |
| Baseline | 1 | (none) | 1 |
| Week 24 | 169 | 2 | 253 |
| Week 48 | 337 | 254 | 421 |
| Week 72 | 505 | 422 | 589 |
| Week 96 | 673 | 590 | 757 |
| Week 120 | 841 | 758 | 925 |
| Week 144 | 1009 | 926 | 1093 |
| Week 168 | 1177 | 1094 | 1261 |
| Week 192 | 1345 | 1262 | 1429 |
| Week 216 | 1513 | 1430 | 1597 |
| Week 240 | 1681 | 1598 | 1765 |
| Week 264 | 1849 | 1766 | 1933 |
| Week 288 | 2017 | 1934 | 2101 |
| Week 312 | 2185 | 2102 | 2269 |
| Week 336 | 2353 | 2270 | 2437 |
| Week 360 | 2521 | 2438 | 2605 |
| Week 384 | 2689 | 2606 | 2773 |
| Week 408 | 2857 | 2774 | 2941 |
| Week 432 | 3025 | 2942 | ≥ 3025 |





## 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Visit Window

Depending on the statistical analysis method, single values may be required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time-to-event analysis would not require 1 value per analysis window.

If multiple valid, nonmissing measurements exist in a postbaseline analysis window, records will be chosen based on the following rules if a single value is needed:

- The record closest to the nominal day for that visit will be selected.
- If there are 2 records that are equidistant from the nominal day, the later record will be selected.
- If there is more than 1 record on the selected day, the average will be taken for continuous data and the worse severity will be taken for categorical data, unless otherwise specified.

#### 3.8.4. Definition of Baseline

Baseline in the LTE is defined as the last nonmissing value on or prior to the first dosing date of study drug in Study GS-US-419-3896, unless specified differently. If there are multiple records with the same time or no time recorded on the same day, the baseline value will be the average of the measurements for continuous data, or the measurement with the lowest severity (eg, normal will be selected over abnormal for safety electrocardiogram [ECG] findings) for categorical data.

#### 4. SUBJECT DISPOSITION

#### 4.1. Subject Enrollment and Disposition

Key study dates (ie, first subject enrolled, last subject enrolled, last subject last visit for the primary endpoint, and last subject last visit for the clinical study report) will be provided.

A summary of subject enrollment will be provided by treatment group for each country, investigator within a country, and overall. The summary will present the number and percentage of subjects enrolled. For each column, the denominator for the percentage calculation will be the total number of subjects analyzed for that column.

A summary of subject disposition will be provided by treatment group. This summary will present the number of subjects in each of the categories listed below:

- All Enrolled Analysis Set
  - By parent study (GS-US-419-4015, GS-US-419-4016, or GS-US-419-3895)
  - By reason for exiting parent study, i.e., either completed to end, due to failure to meet response/remission criteria at W10 or due to protocol-specified disease worsening)
- Safety Analysis Set
- Continuing study drug (for analysis other than the final analysis)
- Completed study drug
- Did not complete study drug with reasons for premature discontinuation of study drug
- Continuing study (for analysis other than the final analysis)
- Completed study
- Did not complete the study with reasons for premature discontinuation of study

For the status of study drug and study completion and reasons for premature discontinuation, the number and percentage of subjects in each category will be provided. The denominator for the percentage calculation will be the total number of subjects in the Safety Analysis Set corresponding to that column.

The following by-subject listings will be provided by subject ID number in ascending order to support the above summary tables:

• Reasons for premature study drug or study discontinuation

• Lot number and kit ID of assigned study medication

## 4.2. Extent of Study Drug Exposure and Adherence

Extent of exposure to study drug will be examined by assessing the total duration of exposure to study drug and the level of adherence relative to the study drug regimen specified in the protocol.

If subjects are continuing study drug at the data cutoff date for an interim analysis, the data cutoff date will be used to impute the last dosing date for the calculation of duration of exposure to study drug and adherence to the study drug.

#### 4.2.1. Duration of Exposure to Study Drug

Total duration of exposure to study drug will be defined as last dosing date minus first dosing date plus 1, regardless of any temporary interruptions in study drug administration, and will be expressed in weeks using up to 1 decimal place (eg, 4.5 weeks). If the last study drug dosing date is missing (for subjects that have stopped treatment or the study as indicated by a study disposition record), the latest date among the treatment (study) disposition date, clinical visit date, laboratory sample collection date, and vital signs assessment date that occurred during the on-treatment period (i.e., after exposure start date) will be used for subjects included in the final analyses or the last available date in the database snapshot at the time of an interim analysis.

If month and year of the last dose are known, and the last study drug dosing date imputed above is different from the month collected, the last date of that month will be used. If only year of the last dose is known, and the last study drug dosing date imputed above is after the year collected, the last date of that year will be used; if the last study drug dosing date imputed above is before the year collected, the first date of that year will be used.

The total duration of exposure to study drug will be summarized using descriptive statistics and using the number (ie, cumulative counts) and percentage of subjects exposed through the following time periods: 1 day, 2 weeks, 4 weeks, 12 weeks, 24 weeks, 36 weeks, 48 weeks, 52 weeks, 60 weeks, and then every 12 weeks from Week 60. Summaries will be provided by treatment group for the Safety Analysis Set.

No formal statistical testing is planned.

#### 4.2.2. Adherence to Study Drug

The total number of tablets taken will be summarized using descriptive statistics.

The presumed total number of tablets taken by a subject will be determined by the data collected on the drug accountability CRF using the following formula:

$$\textit{Total Number of Tablets Taken} = \left(\sum \textit{No.of Tablets Dispensed}\right) - \left(\sum \textit{No.of Tablets Returned}\right)$$

If the bottle was not returned, it is assumed that the subject took all the study drug tablets from the dispensed bottle. The number of tablets returned will be imputed as zero for the given bottle for study drug adherence calculation purposes.

For calculation of the total number of tablets taken for the purposes of interim analyses (ie, prior to the return of all drug bottles), it will be assumed that each subject took the recommended daily dose from the dispensed bottle(s) until either the date of discontinuation, death or data cutoff date (whichever is earliest).

If the bottle has not been returned yet when the interim analysis is conducted, the number of tablets returned will be imputed as total pill count in the dispensed bottle – (the last dosing date – the last bottle dispensed date +1) for the given bottle for study drug adherence calculation purposes.

#### 4.2.2.1. On-Treatment Adherence

The level of on-treatment adherence to the study drug regimen will be determined by the total amount of study drug taken relative to the total amount of study drug expected to be taken during a subject's actual on-treatment period based on the study drug regimen.

The level of on-treatment adherence will be expressed as a percentage using the following formula:

$$On-Treatment\ Adherence\ (\%) = \left(\frac{Total\ Amount\ of\ Study\ Drug\ Taken}{Study\ Drug\ Expected\ to\ be\ Taken\ on\ Treatment}\right)x100$$

Descriptive statistics for the level of on-treatment adherence with the number and percentage of subjects belonging to adherence categories (eg, < 80%,  $\ge 80$  to < 90%,  $\ge 90\%$  to < 120,  $\ge 120$ ) will be provided by treatment group for the Safety Analysis Set.

No formal statistical testing is planned.

A by-subject listing of study drug intake and drug accountability will be provided separately by subject ID number (in ascending order) and visit (in chronological order).

#### 4.3. Protocol Deviations

Subjects who did not meet the eligibility criteria for study entry but enrolled in the study, will be summarized regardless of whether they were exempted by the sponsor or not. The summary will present the number and percentage of subjects who did not meet at least 1 eligibility criterion and the number of subjects who did not meet specific criteria by treatment group based on the All Enrolled Analysis Set. A by-subject listing will be provided for those subjects who did not meet at least 1 eligibility (inclusion or exclusion) criterion. The listing will present the eligibility criterion (or criteria if more than 1 deviation) that subjects did not meet and related comments, if collected.

Protocol deviations occurring after subjects entered the study are documented during routine monitoring. The number and percentage of subjects with important protocol deviations by

deviation category (eg, eligibility criteria, informed consent) will be summarized by treatment group for the All Enrolled Analysis Set. A by-subject listing will be provided for those subjects with important protocol deviations.

# 4.4. Assessment of COVID-19 (Coronavirus Disease 2019) and Ukrainian Conflict Impact

This study was ongoing during the COVID-19 pandemic and the conflict in Ukraine, which have an impact on study conduct. Some subjects were unable to attend onsite visits due to shelter-in-place guidelines, site closures, or other public health measures in response to these situations. This section describes how the impact on study conduct will be handled in the analysis.

#### 4.4.1. Study Drug or Study Discontinuation

Summaries of reasons for discontinuing study drug or study due to COVID-19 will be provided by treatment group and overall, similar to the summary described in the subject enrollment and disposition section (see Section 4.1).

By-subject listing of reasons for premature study drug or study discontinuation due to COVID-19 will be provided if applicable.

#### 4.4.2. Study Drug Interruption

Summaries of number of subjects with study drug interruption due to COVID-19 will be provided by treatment group, if applicable.

By-subject listings of study drug administration for subjects with study drug interruption due to COVID-19 will be provided, if applicable.

#### 4.4.3. Protocol Deviations

Summaries of important protocol deviations due to COVID-19 will be provided, similar to the summary described in the protocol deviations section (Section 4.3).

By-subject listings will be provided for subjects with important protocol deviations related to COVID-19 and the Ukrainian conflict, if applicable.

#### 4.4.4. Missed or Virtual Visits

Summaries of subjects with missed or virtual visits due to the COVID-19 pandemic will be provided for each scheduled study visit by treatment group and overall, for the All Enrolled Analysis Set. For each visit, the summaries will present the number and percentage of subjects who missed the visit due to COVID-19 or had a virtual visit due to COVID-19. For each column, the denominator for the percentage calculation will be the total number of subjects in the All Enrolled Analysis Set for that column.

Overall summaries of the number and percentage of subjects with missed or virtual visits (eg, subjects with at least 1 missed or virtual visit, subjects with 1, 2, 3 or more missed or virtual visits) due to COVID-19 will be provided by treatment group and overall, for the All Enrolled Analysis Set. The denominator for the percentage calculation will be the total number of subjects in the All Enrolled Analysis Set for that column.

By-subject listings of subjects with missed or virtual visits due to COVID-19 will be provided by subject ID number in ascending order.

Information regarding missed or virtual visits due to COVID-19 will be collected as free text in the CRF comment fields. The determination of missed or virtual visits due to COVID-19 will be done using Natural Language Processing (NLP) to search the CRF comment fields. A detailed explanation of the algorithm is given in Appendix 3.

#### 4.4.5. Adverse Events

By-subject listings will be provided for subjects with adverse events of COVID-19, as determined by COVID-19 Standardized MedDRA Query (SMQ) narrow search.

#### 4.4.6. Comments

A by-subject listing of all comments related to the Ukrainian conflict will be provided.

#### 5. BASELINE CHARACTERISTICS

#### 5.1. Demographics and Baseline Characteristics

Subject demographic variables and baseline characteristics below will be summarized by treatment group and overall using descriptive statistics for continuous variables and using number and percentage of subjects for categorical variables. The summary of demographic data will be provided for the Safety Analysis Set. In addition, this summary will be provided for the induction non-responders (see Section 3.4), overall, and by prior exposure to biologic agents.

- Age (years, on the date of the first dose of study drug in Study GS-US-419-3896)
- Age group ( $< 65 \text{ years}, \ge 65 \text{ years}$ )
- Sex at birth (female, male)
- Race
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
- Geographic region (United States [US], non-US)
- Weight (in kg)
- Height (in cm)
- Body mass index (BMI; in kg/m<sup>2</sup>)

A by-subject demographic listing, including the informed consent date, will be provided by subject ID number in ascending order.

#### 5.2. Other Baseline Characteristics

Other baseline characteristics include

- CDAI score
- PRO2 subscores: liquid or very soft stool subscore and abdominal pain subscore
- •
- •
- •
- Concomitant treatment at baseline

- Concomitant use of systemically absorbed corticosteroid and/or immunomodulator, including: a) systemically absorbed corticosteroid only, b) immunomodulator only, c) both, and d) neither
- Prednisone equivalence dose for subjects who are on systemically absorbed corticosteroid (mg/day)
- Prednisone equivalence dose level for subjects who are on systemically absorbed corticosteroid (> 0 to 10 mg/day, > 10 to 20 mg/day, > 20 to 30 mg/day, > 30 mg/day)
- 5-aminosalicylates (yes, no)

These baseline characteristics will be summarized by treatment group and overall using descriptive statistics for continuous variables and using number and percentage of subjects for categorical variables. The summary of these baseline characteristics will be provided for the Safety Analysis Set. In addition, this summary will be provided for the induction non-responders (see Section 3.4), overall, and by prior exposure to biologic agents.

No formal statistical testing is planned.

A by-subject listing of other baseline characteristics will be provided by subject ID number in ascending order.

## 5.3. Medical History

Adverse events which occurred in a parent study and were ongoing when subject took the first dose in this LTE study were recorded as medical history for Study GS-US-419-3896, excluding AEs occurred after Study GS-US-419-3896 informed consent is signed and prior to initiation of Day 1 Study GS-US-419-3896 IMP but related to Study GS-US-419-3896 protocol-mandated procedures.

General medical history data will be collected at enrollment and listed only. General medical history data will be coded using the current version of Medical Dictionary for Regulatory Activities (MedDRA).

#### 6. EFFICACY ANALYSES

#### **6.1.** General Considerations

The efficacy analysis will be conducted on the Safety Analysis Set, defined in Section 3.1.2, unless otherwise specified.

#### 6.1.1. Calculation of CDAI and PRO2 Scores

The CDAI system is a composite index of 8 disease activity variables with scores ranging from 0 to over 600 based upon a composite of symptoms (eg, abdominal pain), signs (the presence of abdominal mass and weight), laboratory values (eg, hematocrit), and physician assessment amongst others. The CDAI has 3 PRO components: liquid or very soft stool frequency, abdominal pain and general wellbeing. The total CDAI score is calculated as a weighted sum of all 8 component subscores. Clinical remission by CDAI is defined as CDAI score < 150 points. If subjects have 1 or more of the 8 component subscores missing, then the subjects will be considered as having insufficient data to determine remission status and their total CDAI score will be considered missing.

The PRO2 instrument has 2 components: liquid or very soft stool frequency subscore and abdominal pain subscore. Clinical remission by PRO2 is defined as an abdominal pain score ≤1 and liquid or very soft stool frequency ≤ 3. If either subscore is missing, the subject will be considered as having insufficient data to determine clinical remission status by PRO2. For further information on the CDAI/PRO2 and calculation rules at baseline and postbaseline, reference is made to Appendix 2.

#### **6.2.** Efficacy Endpoints

#### **6.2.1.** Definition of the Efficacy Endpoints

The secondary endpoints of this study are change in CDAI and PRO2 scores from baseline.

#### 6.2.2. Analysis of the Efficacy Endpoints

#### **CDAI** and **PRO2**

Descriptive statistics and 95% CI based on normal approximation will be used to summarize the absolute values and change from baseline values in CDAI and PRO2 scores by analysis visit and treatment group using observed values. Mean absolute values of each score with 95% CI will be plotted over all analysis visits by treatment group. Mean change from baseline values of each score with 95% CI will also be plotted.







#### 6.5. **Change from Protocol-Specified Efficacy Analyses**

The following are added to the list of efficacy endpoints and the analyses on these endpoints are included as (see Section 6.2.2):

•

#### 7. SAFETY ANALYSES

#### 7.1. Adverse Events and Deaths

#### 7.1.1. Adverse Event Dictionary

Clinical and laboratory AEs will be coded using a recent version of MedDRA. System organ class (SOC), high-level group term (HLGT), high-level term (HLT), preferred term (PT), and lower-level term (LLT) will be provided in the AE dataset.

### 7.1.2. Adverse Event Severity

The severity of AEs was graded using the modified Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. For each episode, the highest grade attained should be reported. If a CTCAE criterion does not exist, the investigator should use the grade or adjectives: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening) or Grade 5 (fatal) to describe the maximum intensity of the adverse event. For purposes of consistency with the CTCAE, these intensity grades are defined in the protocol in Table 7-1 and Appendix 5. The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings. The missing category will be listed last in summary presentation.

#### 7.1.3. Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator selected "Related" on the AE CRF to the question of "Related to Study Treatment." Events for which the investigator did not record relationship to study drug will be considered related to study drug for summary purposes. However, by-subject data listings will show the relationship as missing.

#### 7.1.4. Action Taken With Study Drug

Action taken is recorded for multiple study treatments on the AE CRF. In adverse event summaries a worst-case approach will be applied using all available information. For example, if for at least one of the study treatments "Drug Withdrawn" was recorded, the AE will be categorized as "leading to premature discontinuation of study drug".

#### 7.1.5. Serious Adverse Events

Serious adverse events (SAEs) will be identified and captured as SAEs if the AEs met the definitions of SAEs that were specified in the study protocol. SAEs captured and stored in the clinical database will be reconciled with the SAE safety database before data finalization.

#### 7.1.6. Treatment-Emergent Adverse Events

#### 7.1.6.1. Definition of Treatment-Emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as 1 or both of the following:

- Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug
- Any AEs leading to premature discontinuation of study drug.

#### 7.1.6.2. Incomplete Dates

If the onset date of the AE is incomplete and the AE stop date is not prior to the first dosing date of study drug, then the month and year (or year alone if month is not recorded) of onset determine whether an AE is treatment emergent. The event is considered treatment emergent if both of the following 2 criteria are met:

- The AE onset date is the same as or after the month and year (or year) of the first dosing date of study drug, and
- The AE onset date is the same as or before the month and year (or year) of the date corresponding to 30 days after the date of the last dose of study drug

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date later than the first dosing date of study drug, will be considered to be treatment emergent. In addition, an AE with the onset date missing and incomplete stop date with the same or later month and year (or year alone if month is not recorded) as the first dosing date of study drug will be considered treatment emergent.

#### 7.1.7. Summaries of Adverse Events and Deaths

Treatment-emergent AEs will be summarized based on the Safety Analysis Set.

No formal statistical testing is planned.

### 7.1.7.1. Summaries of AE incidence in Combined Severity Grade Subsets

A brief, high-level summary of the number and percentage of subjects who experienced at least 1 TEAE in the categories described below will be provided by treatment group. All deaths observed in the study will also be included in this summary.

The number and percentage of subjects who experienced at least 1 TEAE will be provided and summarized by SOC, PT, and treatment group. The same summary is provided for the other AE categories described below.

- TEAEs with Grade 3 or higher
- TEAEs with Grade 2 or higher
- Treatment-emergent (TE) treatment-related AEs
- TE treatment-related AEs with Grade 3 or higher
- TE treatment-related AEs with Grade 2 or higher
- TE SAEs
- TE treatment-related SAEs
- TEAEs leading to premature discontinuation of study drug
- TEAEs leading to premature discontinuation of study
- TE AEs leading to death (ie, outcome of death)
- TEAEs leading to temporary interruption of study drug

Multiple events will be counted only once per subject in each summary. Adverse events will be summarized and listed in descending order of frequency, first by SOC, then by PT and then alphabetically. For summaries by severity grade, the most severe grade will be used for those AEs that occurred more than once in an individual subject during the study.

In addition to the above summary tables, the following TEAEs will be summarized by PT only, in descending order of total frequency:

- TEAEs
- TEAEs with Grade 3 or higher
- TE SAEs
- TEAEs leading to premature discontinuation of study drug.

In addition, data listings will be provided for the following:

- All AEs, indicating whether the event is treatment emergent
- All SAEs
- All Deaths
- All SAEs leading to death (ie, outcome of death)

- All AEs with severity of Grade 3 or higher
- All AEs leading to premature discontinuation of study drug
- All AEs leading to premature discontinuation of study
- All AEs leading to temporary interruption of study drug

In addition, an XML file will be created to support EUDRACT reporting for the final analysis containing serious AEs, non-serious AEs and non-serious AEs occurring in at least 5% of subjects in at least one treatment arm, either at system organ class level or at PT level. (This XML file will be created in-house).

#### 7.1.8. Adverse Events of Interest

Adverse events of interest (AEI) include infections, gastrointestinal perforations, herpes zoster, malignancies (excluding non-melanoma skin cancers), non-melanoma skin cancers, major adverse cardiovascular events (MACE), and thromboembolic events. Summaries of the following treatment-emergent AEI will be produced to enhance the analysis of safety data.

- Events of infections presented in the following subcategories:
  - AEs of infections, utilizing all AEs in the MedDRA Infections and Infestations SOC
  - AEs of serious infections, using all AEs in the MedDRA Infections and Infestations SOC that are classified as SAEs
  - AEs of herpes zoster, utilizing an MST list developed by the Sponsor
  - AEs of opportunistic infections, utilizing a narrow scope SMQ
- AEs of malignancies, excluding non-melanoma skin cancers, utilizing an MST list developed by the Sponsor
- AEs of non-melanoma skin cancers, utilizing an MST list developed by the Sponsor
- AEs of gastrointestinal perforation, utilizing an MST list developed by the Sponsor
- AEs of MACE, utilizing a positively adjudicated event list, presented in the following subcategories (Section 7.1.8.1):
  - Cardiovascular (CV) death
  - Non-fatal myocardial infarction (MI)
  - Non-fatal stroke
- AEs of arterial systemic thromboembolism (ASTE), utilizing a positively adjudicated event list (Section 7.1.8.1)

- AEs of venous thromboembolism (VTE), utilizing a positively adjudicated event list, presented in the following subcategories (Section 7.1.8.1):
  - Venous Thrombotic and Embolic Events
  - Other

The number and percentage of subjects with a reported event will be summarized for each treatment group by PT for each AEI category. Data listings for AEI will also be provided.

A by-subject listing for subjects with potential events for adjudication (MACE, ASTE, and VTE) and their respective adjudication results will be provided.

A by-subject listing of thromboembolic history and risk factors will be provided for subjects with potential events for adjudication (MACE, ASTE, and VTE).

#### 7.1.8.1. Cardiovascular Safety Endpoint Adjudication Committee

An independent cardiovascular safety endpoint adjudication committee (CVEAC) was formed to periodically review and adjudicate all potential MACE and thromboembolic events in a blinded manner. To identify potential MACE and thromboembolic events, the following AEs were sent for adjudication. Refer to the Cardiovascular Event Adjudication Charter for more details.

- All AEs leading to death
- CV events (meeting seriousness criteria), utilizing an MST list developed by the Sponsor
- MI, utilizing a narrow scope SMQ
- Unstable angina (meeting hospitalization criteria), utilizing an MST list developed by the Sponsor
- Transient ischemic attack, utilizing an MST list developed by the Sponsor
- Stroke, utilizing an MST list developed by the Sponsor
- Cardiac failure (meeting hospitalization criteria), utilizing an MST list developed by the Sponsor
- Percutaneous coronary intervention, utilizing an MST list developed by the Sponsor
- Embolic and thrombotic events, utilizing a narrow scope SMQ

The CVEAC will review the above AEs, and related clinical data to adjudicate whether the criteria for MACE (CV death, MI, and/or stroke), ASTE, and VTE have been met for each AE.

## 7.2. Laboratory Evaluations

Laboratory data collected during the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries of laboratory data will be provided for the Safety Analysis Set and will include data collected up to the last dose of study drug plus 30 days for subjects who have permanently discontinued study drug, or all available data at the time of the database snapshot for subjects who were ongoing at the time of an interim analysis. The analysis will be based on values reported in conventional units. When values are below the LOQ, they will be listed as such, and the closest imputed value will be used for the purpose of calculating summary statistics as specified in Section 3.7. Hemolized test results will not be included in the analysis, but they will be listed in by-subject laboratory listings.

A by-subject listing for laboratory test results will be provided by subject ID number and time point in chronological order for hematology, serum chemistry, urinalysis, lipid profile, and serum immunoglobulin separately. Values falling outside of the relevant reference range and/or having a severity grade of 1 or higher on the CTCAE severity grade will be flagged in the data listings, as appropriate.

Hematocrit results collected from local laboratories due to COVID-19 impact will not be included in the safety laboratory summary, but will be included in the listing with a flag to indicate which records were collected at local laboratories.

No formal statistical testing is planned.

### 7.2.1. Summaries of Numeric Laboratory Results

Descriptive statistics will be provided by treatment group for each laboratory test specified in the study protocol within hematology and chemistry panels including creatinine clearance, and also laboratory tests from lipids panel (under fasting status) including total cholesterol, LDL, HDL, triglycerides, non-HDL cholesterol (total cholesterol minus HDL cholesterol), LDL/HDL ratio, and total immunoglobulin (Ig), IgA, IgM, and IgG, as follows:

- Baseline values
- Values at each postbaseline time point
- Change from baseline at each postbaseline time point

A baseline laboratory value will be defined as the last measurement obtained on or prior to the date/time of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the visit value minus the baseline value. The mean, median, Q1, Q3, minimum, and maximum values will be displayed to the reported number of digits; SD values will be displayed to the reported number of digits plus 1.

Median (Q1, Q3) of the observed change from baseline values for aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, alkaline phosphatase, serum creatine, creatinine clearance, creatine phosphokinase, white blood cell count, absolute neutrophils,

absolute lymphocytes, hemoglobin, platelets, total cholesterol, LDL, HDL, total Ig, IgG, IgA, and IgM, will be plotted using a line plot by treatment group and time point.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3.

#### 7.2.2. Graded Laboratory Values

The CTCAE Version 4.03 will be used to assign toxicity grades (0 to 4) to laboratory results for analysis. Grade 0 includes all values that do not meet the criteria for an abnormality of at least Grade 1. For laboratory tests with criteria for both increased and decreased levels, analyses for each direction (ie, increased, decreased) will be presented separately.

#### 7.2.2.1. Treatment-Emergent Laboratory Abnormalities

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days for subjects who permanently discontinued study drug, or the last available date in the database snapshot for subjects who were still on treatment at the time of an interim analysis. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment emergent.

## 7.2.2.2. Treatment-Emergent Marked Laboratory Abnormalities

Treatment-emergent marked laboratory abnormalities are defined as values that increase from baseline by at least 3 toxicity grades at any postbaseline time point, up to and including the date of the last dose of study drug plus 30 days for subjects who permanently discontinued study drug or the last available date in the database snapshot for subjects who were still on treatment at the time of an interim analysis. If the relevant baseline laboratory value is missing, any Grade 3 or 4 values observed within the timeframe specified above will be considered treatment-emergent marked abnormalities.

#### 7.2.2.3. Summaries of Laboratory Abnormalities

The following summaries (number and percentage of subjects) for treatment-emergent laboratory abnormalities will be provided by lab test and treatment group; subjects will be categorized according to the most severe postbaseline abnormality grade for a given lab test:

- Graded laboratory abnormalities
- Grade 3 or 4 laboratory abnormalities
- Marked laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of subjects with nonmissing postbaseline values up to 30 days after last dosing date.

A by-subject listing of treatment-emergent Grade 3 or 4 laboratory abnormalities will be provided by subject ID number and time point in chronological order. This listing will include all test results that were collected throughout the study for the lab test of interest, with all applicable severity grades displayed.

#### 7.2.3. Liver-Related Laboratory Evaluations

Liver-related abnormalities after initial study drug dosing will be examined and summarized using the number and percentage of subjects who were reported to have the following laboratory test values for postbaseline measurements:

- Aspartate aminotransferase (AST): (a) > 3 times of the upper limit of normal (ULN) reference range; (b) > 5 × ULN; (c) > 10 × ULN; (d) > 20 × ULN
- Alanine aminotransferase (ALT): (a) > 3 × ULN; (b) > 5 × ULN; (c) > 10 × ULN;
   (d) > 20 × ULN
- AST or ALT  $> 3 \times ULN$  and total bilirubin  $> 2 \times ULN$

The summary will include data from all postbaseline visits up to 30 days after the last dose of study drug. For individual laboratory tests, subjects will be counted once based on the most severe postbaseline values. For both the composite endpoint of AST or ALT and total bilirubin, subjects will be counted once when the criteria are met at the same postbaseline visit date. The denominator is the number of subjects in the Safety Analysis Set who have nonmissing postbaseline values of all relevant tests at the same postbaseline visit date. A listing of subjects who met at least 1 of the above criteria will be provided.

#### 7.3. Body Weight and Vital Signs

Descriptive statistics will be provided by treatment group for body weight, BMI and vital signs (resting blood pressure [systolic blood pressure and diastolic blood pressure], respiratory rate, pulse and temperate) as follows:

- Baseline value
- Values at each postbaseline time point
- Change from baseline at each postbaseline time point

A baseline value will be defined as the last available value collected on or prior to the date/time of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the postbaseline value minus the baseline value. Body weight and vital signs measured at unscheduled visits will be included for the baseline value selection.
In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3. No formal statistical testing is planned.

A by-subject listing of vital signs will be provided by subject ID number and time point in chronological order. Body weight, height, and BMI will be included in the vital signs listing, if space permits. If not, they will be provided separately.

Body weight results measured by subjects at home from virtual visits due to COVID-19 impact will not be included in the vital signs summary, but will be included in the listing with a flag to indicate which records were collected at home.

#### 7.4. Concomitant Medications

Medications collected during the study will be coded using the current version of the World Health Organization (WHO) Drug dictionary.

Concomitant medications are defined as medications taken while a subject took study drug. Use of concomitant medications will be summarized by therapeutic subgroup (ATC level 2) and preferred name using the number and percentage of subjects for each treatment group. A subject reporting the same medication more than once will be counted only once when calculating the number and percentage of subjects who received that medication. The summary will be ordered in descending overall frequency, first by ATC class and then by preferred term. For drugs with the same frequency, sorting will be done alphabetically.

For the purposes of analysis, any medications with a start date prior to or on the first dosing date of study drug and continued to be taken after the first dosing date, or started after the first dosing date but prior to or on the last dosing date of study drug will be considered concomitant medications. Medications started and stopped on the same day as the first dosing date or the last dosing date of study drug will also be considered concomitant. Medications with a stop date prior to the date of first dosing date of study drug or a start date after the last dosing date of study drug will be excluded from the concomitant medication summary. If a partial stop date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) prior to the date of first study drug administration will be excluded from the concomitant medication summary. If a partial start date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) after the study drug stop date will be excluded from the concomitant medication summary. Medications with completely missing start and stop dates will be included in the concomitant medication summary, unless otherwise specified. Summaries will be based on the Safety Analysis Set. No formal statistical testing is planned.

All concomitant medications (other than per-protocol study drugs) will be provided in a by-subject listing sorted by subject ID number and administration date in chronological order.

#### 7.5. Electrocardiogram Results

A frequency table of the investigators' assessment of ECG results at each visit will be presented by treatment group, using the following categories: normal; abnormal, not clinically significant; abnormal, clinically significant. The number and percentage of subjects in each classification group will be presented.

No formal statistical testing is planned.

A by-subject listing for ECG assessment results will be provided by subject ID number and time point in chronological order.

#### 7.6. Other Safety Measures

A data listing will be provided for subjects who become pregnant during the study.

| l |
|---|

#### 9. SOFTWARE

SAS® Software Version 9.4. SAS Institute Inc., Cary, NC, USA.

#### 10. SAP REVISION

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|
| Original Gilead draft<br>(11 February 2022) | | | |
| Draft 0.3<br>(11 July 2022) | Global | Editorial changes have been made throughout the SAP, where appropriate | To align with GLPG wording / template |
| | 4.4 | Added assessment of Ukrainian conflict impact | To better understand the Ukrainian conflict impact on subject disposition and missing data |
| | 6.2 | Added remission by CDAI and PRO2 as efficacy endpoints | To support the secondary endpoints. |
| | 6.3, 7.1.8 | Added subgroup analyses for efficacy endpoints and adverse events | To assess benefit/risk in subjects who completed the parent study and subjects who met protocol-specified efficacy discontinuation criteria |
| Draft 0.4<br>(1 Augustus 2022) | Global | Editorial changes have been made throughout the SAP, where appropriate | For clarification, based on team feedback |
| | 5.2 | Added baseline disease characteristics by subgroup | To complement the efficacy/safety subgroup analyses |
| | 7.1.6 | AEs will be presented ordered by total frequency, not alphabetically | Requested by medical writing |
| | 7.5 | Addition of ECG shift table | Requested by medical leads |
| Draft 0.5<br>(12 November 2022) | Global | Clarifications and corrections have been made throughout the SAP, where appropriate | Based on dry-run findings |
| | 3.4 | Update definition subgroups. | Based on internal discussion |
| | 4.4.5 | Replacing COVID impact indicator by listing of AEs related to COVID | The impact indicator is a Gilead-defined analysis. Not deemed valuable |
| | 7.4 | Addition of ATC level 2 in summaries of concomitant medications | Requested by medical leads |
| | 7.5 | ECG shift table replaced by frequency table | Baseline ECG not available in this study |
| | Title page | Update medical leader | |

| Final Version 1.0<br>(13 January 2023) | 4.4 | Reduction of planned analyses related to the impact of the Ukrainian conflict | Data availability |
|---|---|---|---|
| | 5.2 | Update prednisone dose categories | Requested by medical leads |
| | 7.1.4 | Added section on the handling of<br>"action taken" information in the<br>summaries of AEs | Clarification |
| | Appendix 5 | Addition of MST lists based on the latest MedDRA version | For transparency on which lists were used at the time of analysis |
| Final Version 2.0<br>(1 August 2023) | 3.2, 3.4, 5.1,<br>5.2, 6.3 | Extension of analyses of baseline characteristics and efficacy endpoints in the subset of induction non-responders: by prior exposure, addition of imputation rules | For better understanding of this specific subgroup |
| | 7.1.7 | Removal of specific AE summaries | Considered unnecessary by the team |
| | 7.1.8 | Addition of subcategories VTE | Request medical safety |
| | 7.1.9 | Removal of subgroup analyses for AE | Considered unnecessary by the team |
| | 7.2.2 | Removal lab shift tables | Considered unnecessary by the team |

#### 11. APPENDICES

| Appendix 1. | Schedule of Assessments | 44 |
|-------------|-------------------------------------|----|
| * * | CDAI and PRO2 Calculation | |
| * * | Data Collection of COVID-19 Data | |
| * * | Calculation of Standard Body Weight | |
| * * | MST Lists for AEs of Interest | |

#### **Appendix 1.** Schedule of Assessments

| | Day 1ª | Week 2 | Week 4 | Every<br>4 Weeks<br>from<br>Day 1 | Week 12 and<br>then every<br>12 Weeks<br>from Day 1<br>Clinic Visit | Every 24 Weeks from Day 1 Clinic Visit | Every<br>48 Weeks<br>from<br>Day 1<br>Clinic<br>Visit | Early<br>Termination<br>(ET) Visit | Post-Treatment (PTx) <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|
| <b>Study Procedures</b> | | ± 3 days | ± 3 days | ±7 days | ±7 days | ± 7 days | ±7 days | | ± 3 days |
| Written Informed Consent | X | | | | | | | | |
| Review Inclusion/Exclusion<br>Criteria | X | | | | | | | | |
| Medical History | X | | | | | | | | |
| Symptom-Directed Examination (as needed) | | | | | X | | | X | X |
| Perianal fistulae assessment<br>(for subjects rolling over from<br>GS-US-419-4016 <b>only</b> ) ° | | | | | X | | | X | X |
| Vital Signs <sup>d</sup> | X | X | X | | X | | | X | X |
| Height | X | | | | | | | | |
| Weight | X | X | X | | X | | | X | X |
| Hematology | X | X | X | | X | | | X | X |
| Chemistry | X | X | X | | X | | | X | X |
| Lipid Profile (fasting) <sup>e</sup> | | | | | | X | | | |
| Urinalysis | X | | | | | X | | | |
| Pregnancy Test <sup>f</sup> | X | | X | X | | | | X | X |
| HBV DNA monitoring (Japan) <sup>g</sup> | X | | X | X | | | | | |
| HBV DNA monitoring (other regions) <sup>h</sup> | X | | | | X | | | | |
| TB Assessment <sup>i</sup> | X | | | | | | X | | |

| | Day 1ª | Week 2 | Week 4 | Every<br>4 Weeks<br>from<br>Day 1 | Week 12 and<br>then every<br>12 Weeks<br>from Day 1<br>Clinic Visit | Every<br>24 Weeks<br>from<br>Day 1<br>Clinic<br>Visit | Every<br>48 Weeks<br>from<br>Day 1<br>Clinic<br>Visit | Early<br>Termination<br>(ET) Visit | Post-Treatment<br>(PTx) <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|
| Study Procedures | | ± 3 days | ± 3 days | ±7 days | ±7 days | ±7 days | ±7 days | | ± 3 days |
| 12-lead ECG | | | | | | | X | | |
| Serum immunoglobulin | X | | | | | | | | |
| e-Diary Instruction & Review <sup>1</sup> | X | X | X | | X | | | | |
| PRO2 <sup>m</sup> | X | X | X | | X | | | X | |
| CDAI <sup>m</sup> | X | X | X | | X | | | X | |
| Enrollment | X | | | | | | | | |
| Study Drug Dispensation | X | | X | | X | | | | |
| Adverse Events <sup>o</sup> | X | X | X | | X | | | X | X |
| Concomitant Medications | X | X | X | | X | | | X | X |

a Day 1 visit for this study may occur at the same time as the final scheduled treatment visit of the prior filgotinib study. All procedures necessary for the final visit in the prior filgotinib study will be completed as well as any additional procedures required for this study. Procedures that are duplicates of the final visit from prior filgotinib study do

k

- not need to be performed again for this protocol. Day 1 may be delayed up to 10 days. If Day 1 of LTE is not the same as the last study visit of the prior study, a full set of Day 1 procedures should be performed. If a subject has already taken study drug for that day within the parent protocol, first dose should take place on Day 2.
- b The Post-Treatment (PTx) Visit should occur 30 days after the last dose of study drug.
- c The perianal fistula assessment entails tracking the clinical status of draining external openings of perianal fistulae that were identified at baseline of Study GS-US-419-4016. For additional details on the perianal assessment, refer to the Perianal Fistula Assessment Manual
- d Vital signs include resting blood pressure, respiratory rate, pulse, and temperature.
- e Fasting means no food or drink except water, for 8 hours
- f Females who are of childbearing potential only. A urine pregnancy test must be completed in clinic every 4 weeks at a minimum. If any pregnancy test is positive, study drug should be immediately interrupted and the subject should have a serum pregnancy test in clinic.
- g In Japan, subjects with negative HBsAg, positive HBcAb and/or positive HBsAb in a parent CD protocol require HBv DNA monitoring every 4 weeks in accordance with local guidelines (Protocol Section 6.2.1).
- h In other regions, subjects with negative HBsAg and positive HBcAb require HBV DNA monitoring every 3 months in accordance with local guidelines (Protocol Section 6.2.1)
- i Subjects who were previously treated for TB do not need to have yearly QuantiFERON® (or centrally reported equivalent assay) tests but should be screened at least yearly for signs and symptoms of reactivation.
- At Day 1 visit, review diary of subject reported components from parent study. Subjects should begin filling out the Diary on Day 1 visit and continue to fill it out throughout the study.
- m Colonoscopy with biopsies is optional per standard of care. The date of the procedure may be requested for accuracy of data analysis.
- o Ongoing AEs from previous filgotinib studies should be recorded as medical history. Collection of AEs and SAEs related to protocol-mandated procedures will begin once informed consent is signed and will continue through the Post-Treatment (PTx) Visit.

#### **Appendix 2. CDAI and PRO2 Calculation**

The total CDAI score is a weighted sum of all 8 variables as specified in Table 11-1, and the PRO2 scores will be assessed according to Table 11-2. Details for the calculations of CDAI and PRO2 scores at baseline and post-baseline visits are provided in this appendix.

Table 11-1. Calculation of Total CDAI Score

| Variable no. | Variable | Variable description | Multiplier |
|---|---|---|---|
| 1 | Liquid or very soft stool | Daily stool count is summed for 7 days | 2 |
| 2 | Abdominal pain | Sum of 7 days of daily ratings as 0 = none, 1 = mild, 2 = moderate, 3 = severe | 5 |
| 3 | General wellbeing | Sum of 7 days of daily ratings as<br>0 = generally well, 1 = slightly below par,<br>2 = poor, 3 = very poor, 4 = terrible | 7 |
| 4 | Complications | Number of listed complications: - Arthritis or arthralgia - Erythema nodosum, pyoderma gangrenosum or apthous stomatitis - Iritis or uveitis - Anal fissures or fistulae or abscess - Other fistula - Fever over 37.8 C [100 F] during past week | 20 each |
| 5 | Use of anti-diarrheal medications | Use of diphenoxylate or loperamide or other opiate for diarrhea $0 = \text{No}, 1 = \text{Yes}$ | 30 |
| 6 | Abdominal mass | 0 = none, 2 = questionable, 5 = definite | 10 |
| 7 | Hematocrit* | Males: 47 – Hct [%] Females: 42 – Hct [%] *Result must be greater than or equal to 0. If negative result enter 0 | 6 × difference |
| 8 | Weight* | Percentage deviation from standard weight (1 – weight / standard weight) × 100 *Limit of -10 (Result must be greater than or equal to -10) | 1 |
| CDAI score | | | TOTAL |

CDAI = Crohn's Disease Activity Index; Hct = hematocrit

| <b>Table 11-2.</b> | Calculation of PRO2 Components |
|--------------------|--------------------------------|
|--------------------|--------------------------------|

| Variable no. | Variable | Variable Description |
|---|---|---|
| 1 | Liquid or very soft stool | Mean of the daily (liquid or very soft) stool count for 7 days |
| 2 | Abdominal pain | <b>Mean</b> of 7 days of daily ratings as 0 = none, 1 = mild, 2 = moderate, 3 = severe |

Each PRO2 subscore will be rounded to the nearest integer (eg, 2) in the determination of subject eligibility for the study and calculation of endpoints.

The 3 patient-reported outcome components for CDAI (and each subscore for PRO2) are determined using an electronic daily diary, which collects subject reported components directly. Given that the ileocolonoscopy procedure (non-protocol-directed procedures) may impact the validity of the diary data, diary data collected 1 day prior to and on the day of the procedure will not be used in the calculation of CDAI and PRO2 subscores for all visits. Those days are called non-evaluable days.

#### Calculation of CDAI and PRO2 Scores for Baseline and Post-baseline Visits

The calculations of CDAI and PRO2 scores for baseline and post-baseline visits are specified below:

- 1) The Day 1 visit date will be used as the anchor day for baseline and following visit dates will be used as the anchor day for post-baseline visits. The visit date for each analysis visit will be selected as the anchor day among all scheduled visits and unscheduled visits where CDAI were assessed within the analysis window as defined in Section 3.8.2. Only diary data collected on evaluable days within a 10-day window which starts 10 days prior to the selected visit date (V-Day 1) and ends on the day prior to V-Day 1 will be used for calculation.
- 2) If there are 7 or more evaluable records within the 10-day window, take the **sum** of the 7 evaluable records closest to V-Day 1 for the corresponding CDAI subject-reported component. For the corresponding PRO2 component, take the **average** of the 7 evaluable records within the 10-day window closest to V-Day 1.
  - a) If there are 4 or more (but less than 7) evaluable records within this 10-day window, the average of the available records will be taken, and then multiplied by 7 for the corresponding CDAI patient-reported component. For the corresponding PRO2 component, the average of the available records will be taken.
  - b) If subjects do not have at least 4 evaluable records within this 10-day window, the corresponding CDAI patient-reported component, and the corresponding PRO2 component will not be calculated and will be considered as missing for that visit.

A schema of this approach and some examples are included below for further explanation:

Figure 1. Selection of Diary Data for the Calculation for Baseline and Postbaseline Visits



Table 11-3. Calculation of CDAI Patient-Reported Outcome Components and PRO2 Scores for Baseline and Post-baseline Visits

| | Diary Day Looking Backwards from Visit<br>Date (V-Day) | | | | | | | | Days for<br>Calculation | Sum of 7 Days<br>(CDAI<br>Patient-Reported<br>Component) | Average<br>of<br>7 Days<br>(PRO2) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Example | -10 | -9 | -8 | -7 | -6 | -5 | -4 | -3 | -2 | -1 | | | |
| Diary<br>Subscore<br>1 | 1 | 2 | 2 | M | 0 | 1 | 2 | 2 | 1 | x | -2,-3,-4,-5,-6,-<br>8,-9 | 10.0 | 1.4 |
| Diary<br>Subscore<br>2 | M | M | 1 | M | x | IL | 2 | 2 | 1 | М | -2,-3,-4, -8 | 10.5 | 1.5 |
| Diary<br>Subscore<br>3 | M | M | 1 | x | IL | M | M | 2 | 1 | М | -2,-3,-8 | Missing | Missing |
| Diary<br>Subscore<br>4 | 0 | M | 2 | 2 | 1 | 0 | M | 2 | X | IL | -3,-5,-6,-7,-8,-<br>10 | 8.2 | 1.2 |

M = Missing; IL = Ileocolonoscopy day; X = non-evaluable (due to preparation for ileocolonoscopy).

Days are named relative to visit date (V-Day 1), where V-Day -1 is the day prior to V-Day 1.

Rounding of subscores into one decimal place is for displaying purpose only. When calculating the total CDAI scores, the subscores will not be rounded.

3) The CDAI total score for a specific visit is based on a weighted sum (rounded to the nearest integer) of all 8 components. The CDAI total score will be set to 0 in the case the calculation leads to a CDAI total score < 0. Each component will be selected within the analysis window as defined in Table 3-1 in Section 3.8.2.

If subjects have at least 1 of the 8 CDAI components missing, then their total CDAI score will be considered missing. If at least 1 out of the 6 complications under the complication component is missing, then the complication component will be considered missing.

CONFIDENTIAL

4) The PRO2 subscores for a specific visit are based on the evaluation of liquid or very soft stool frequency and abdominal pain subscores individually (rounded to the nearest integer) within the analysis window as defined in Section 3.8.2.

#### Source of Information Used for CDAI and PRO2 Calculation

The sources of information used for the calculations of CDAI and PRO2 scores as described above are given in  (the calculated scores from ERT data w ill not be used for data analysis). Hematocrit results collected from local laboratories and body weight measured at home due to COVID-19 impact will be used in CDAI calculation.

**Table 11-4.** Sources of Information for Calculating CDAI and PRO2 Scores

| Variable in Calculation | Data Source |
|---|---|
| Visit Date | VISITDAT in VISDT dataset from eCRF data |
| Stool Frequency Diary Data | QSSTRESN in DIARY dataset with QSTESTCD="SOFSTOOL" from vendor ERT data |
| Abdominal Pain Diary Data | QSSTRESN in DIARY dataset with QSTESTCD="ABDPAIN" from vendor ERT data |
| Subject Standard Weight | SEX_STD in DM dataset and HEIGHT_STD in VSPERF dataset from eCRF data will be used to determine the standard weight based on Appendix 4. |
| Subject Actual Weight | WEIGHT_STD in VSPERF dataset from eCRF data |
| Hematocrit Value | CNVRESN in COVLAB dataset with LBTEST="Hematocrit" from vendor Covance data or LBORRES in LB_HEM dataset with LBTEST="Hematocrit" from eCRF data if collected in local laboratory due to COVID-19 impact |

Note: eCRF = electronic case report form(s). ERT is the vendor that electronically collects patient and investigator reported outcomes.

#### **Appendix 3.** Data Collection of COVID-19 Data

This appendix describes the clinical trial site collection of COVID-19 data pertaining to missed/virtual visits and the data processing algorithm that will be used to determine which visits are missing and which visits are virtual.

#### **Data Collection**

A COVID-19 supplement to the eCRF Completion Guidelines (CCG) was provided by Clinical Data Management to instruct clinical trial sites with data entry expectations pertaining to scenarios related to the COVID-19 pandemic. If a visit was missed, sites were instructed to enter "Visit missed due to COVID-19" and if an in-person visit was conducted virtually, sites were instructed to enter "Virtual visit due to COVID-19".

#### **Determination of Missed and Virtual Visits**

Natural Language Processing (NLP) will be used to search the CRF comment fields to identify instances of "COVID-19", "Virtual", or synonyms (see Table 11-5). The search terms will be maintained in a global lookup table and can be modified to tune the NLP model. Any comments with COVID-19 search terms, "Missed visit" or "Virtual visit will be assigned as follows:

- i. If COVID-19 terms are identified through NLP and the visit date is missing, then result is "Missed Visit"
- ii. If COVID-19 and Virtual terms are identified through NLP for a visit, then result is "Virtual Visit". When there are multiple records for the same subject and the same visit, if one record could be categorized as "Virtual Visit", all records associated with this subject and this visit will be categorized as "Virtual Visit"
- iii. Otherwise result is missing

Table 11-5. Example Search Terms for "COVID-19" and "Virtual" Used to Identify Missed/Virtual Visits

| Search Terms for "COVID-19" | Search Terms for "Virtual" |
|-----------------------------|----------------------------|
| COVID19 | VIRTUAL |
| CORONA | TELEMED |
| CORONAVIRUS | TELEHEALTH |
| PANDEMIC | TELEPHONE |
| OUTBREAK | REMOTE |
| CRISIS | TELEMEDICINE |
| LOCKDOWN | TELECONSULTATION |
| QUARANTINE | TELEPHONICALLY |
| SHELTER | PHONE |
| | HOME VISIT |
| | ZOOM |
| | SKYPE |

#### Appendix 4. Calculation of Standard Body Weight

The following table will be used to determine the standard body weight for each subject. Height from the eCRF will be used and is assumed to be measured without shoes.

| Women | | | |
|---|---|---|---|
| Height in <i>cm</i> (in shoes)* | Standard Weight<br>in <i>kg</i> | Height in <i>cm</i><br>(in shoes)* | Standard Weight<br>in <i>kg</i> |
| 127 | 41.2 | 163 | 60.2 |
| 128 | 41.7 | 164 | 60.7 |
| 129 | 42.3 | 165 | 61.3 |
| 130 | 42.8 | 166 | 61.9 |
| 131 | 43.3 | 167 | 62.4 |
| 132 | 43.8 | 168 | 62.9 |
| 133 | 44.4 | 169 | 63.4 |
| 134 | 44.9 | 170 | 63.9 |
| 135 | 45.4 | 171 | 64.5 |
| 136 | 45.9 | 172 | 65.0 |
| 137 | 46.4 | 173 | 65.5 |
| 138 | 47.0 | 174 | 66.0 |
| 139 | 47.5 | 175 | 66.6 |
| 140 | 48.0 | 176 | 67.2 |
| 141 | 48.6 | 177 | 67.7 |
| 142 | 49.1 | 178 | 68.3 |
| 143 | 49.6 | 179 | 68.8 |
| 144 | 50.2 | 180 | 69.3 |
| 145 | 50.7 | 181 | 69.8 |
| 146 | 51.2 | 182 | 70.3 |
| 147 | 51.8 | 183 | 70.8 |
| 148 | 52.3 | 184 | 71.3 |
| 149 | 52.8 | 185 | 71.8 |
| 150 | 53.1 | 186 | 72.3 |
| 151 | 54.1 | 187 | 72.8 |
| 152 | 54.5 | 188 | 73.3 |
| 153 | 55.0 | 189 | 73.8 |
| 154 | 55.4 | 190 | 74.3 |
| 155 | 55.9 | 191 | 74.9 |
| 156 | 56.4 | 192 | 75.4 |
| 157 | 57.0 | 193 | 76.0 |
| 158 | 57.5 | 194 | 76.5 |
| 159 | 58.1 | 195 | 77.0 |
| 160 | 58.6 | 196 | 77.6 |
| 161 | 59.1 | 197 | 78.1 |
| 162 | 59.6 | 198 | 78.6 |

<sup>\*</sup> add 2.0 cm if shoeless. Please round height to a whole number and select the appropriate standard weight (eg, height 157.4 cm will be rounded to 157 cm; 157.5 cm will be rounded to 158 cm.)

| Men | | | |
|---|---|---|---|
| Height in <i>cm</i> (in shoes)* | Standard Weight<br>in <i>kg</i> | Height in <i>cm</i> (in shoes)* | Standard Weight<br>in <i>kg</i> |
| 142 | 54.4 | 179 | 71.9 |
| 143 | 54.9 | 180 | 72.4 |
| 144 | 55.4 | 181 | 73.0 |
| 145 | 55.8 | 182 | 73.6 |
| 146 | 56.3 | 183 | 74.3 |
| 147 | 56.8 | 184 | 74.8 |
| 148 | 57.2 | 185 | 75.5 |
| 149 | 57.7 | 186 | 76.2 |
| 150 | 58.2 | 187 | 76.9 |
| 151 | 58.6 | 188 | 77.6 |
| 152 | 59.1 | 189 | 78.2 |
| 153 | 59.6 | 190 | 78.8 |
| 154 | 60.0 | 191 | 79.6 |
| 155 | 60.5 | 192 | 80.4 |
| 156 | 61.0 | 193 | 81.2 |
| 157 | 61.4 | 194 | 82.1 |
| 158 | 61.9 | 195 | 82.9 |
| 159 | 62.2 | 196 | 83.8 |
| 160 | 62.6 | 197 | 84.7 |
| 161 | 62.9 | 198 | 85.4 |
| 162 | 63.3 | 199 | 86.1 |
| 163 | 63.7 | 200 | 86.7 |
| 164 | 64.1 | 201 | 87.4 |
| 165 | 64.6 | 202 | 88.0 |
| 166 | 65.0 | 203 | 88.8 |
| 167 | 65.5 | 204 | 89.4 |
| 168 | 66.0 | 205 | 90.1 |
| 169 | 66.6 | 206 | 90.7 |
| 170 | 67.1 | 207 | 91.4 |
| 171 | 67.6 | 208 | 92.1 |
| 172 | 68.1 | 209 | 92.7 |
| 173 | 68.7 | 210 | 93.4 |
| 174 | 69.2 | 211 | 94.1 |
| 175 | 69.7 | 212 | 94.8 |
| 176 | 70.3 | 213 | 95.5 |
| 177 | 70.8 | 214 | 96.1 |
| 178 | 71.3 | | |

<sup>\*</sup> add 2.0 cm if shoeless. Please round height to a whole number and select the appropriate standard weight (eg, height 157.4 cm will be rounded to 157 cm; 157.5 cm will be rounded to 158 cm.)

#### **MST Lists for AEs of Interest**

#### Herpes Zoster - Galapagos Search Term List MedDRA Version 25.0


22323

## Malignancies, Excluding Nonmelanoma Skin Cancers - Galapagos Search Term List MedDRA Version 25.0


## Nonmelanoma Skin Cancers - Galapagos Search Term List MedDRA Version 25.0


# Gastrointestinal Perforations - Galapagos Search Term List MedDRA Version 25.0


## Unstable Angina - Galapagos Search Term List MedDRA Version 25.0


## Transient Ischemic Attack - Galapagos Search Term List MedDRA Version 25.0


# Transient Ischemic Attack - Galapagos Search Term List MedDRA Version 25.0


Stroke - Galapagos Search Term List MedDRA Version 25.0


Stroke - Galapagos Search Term List MedDRA Version 25.0


## Cardiac Failure - Galapagos Search Term List MedDRA Version 25.0


### Cardiac Failure - Galapagos Search Term List MedDRA Version 25.0


# Percutaneous Coronary Intervention - Galapagos Search Term List MedDRA Version 25.0


## Percutaneous Coronary Intervention - Galapagos Search Term List MedDRA Version 25.0


## Percutaneous Coronary Intervention - Galapagos Search Term List MedDRA Version 25.0


Specific AE directly associated with the pathogen causing COVID-19 - Galapagos Search Term List MedDRA Version 25.0  $\,$ 


### Signature Page for gs-us-419-3896-sap 22323



Signature Page for gs-us-419-3896-sap43952\_42958\_121886